CLINICAL TRIAL: NCT00120835
Title: An Open-Label, Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and the Antiviral Activity of NM283 When Administered Alone and in Combination With Pegylated Interferon Alfa 2b to Treatment-Naive Adults With Genotype-1 Chronic Hepatitis C
Brief Title: Valopicitabine When Administered Alone and in Combination With Interferon to Treatment-Naive Patients With Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV-08A-003
Record Dates: First submitted 2005-07-11; First posted 2005-07-19 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis C
Keywords: Genotype-1; Treatment-Naive
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — valopicitabine

INTERVENTIONS:
Drug: valopicitabine
Drug: pegylated interferon

SUMMARY:
This study is being conducted in treatment-naive patients (no previous hepatitis C treatment) to evaluate the safety of valopicitabine (NM283) alone and together with pegylated interferon, a drug approved by the Food and Drug Administration for the treatment of hepatitis C infection. This study is also evaluating the ability of valopicitabine to decrease the amount of hepatitis C virus in the body. The results for patients taking valopicitabine alone will be compared with the results for patients taking valopicitabine together with pegylated interferon.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history compatible with genotype-1, chronic hepatitis C infection
* Treatment-naive (patient has received no previous therapy for hepatitis C viral infection)

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant
* Patient is co-infected with hepatitis B or HIV

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-07

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Bradenton, Florida
  - San Antonio, Texas
- Santurce, Puerto Rico